CLINICAL TRIAL: NCT03129555
Title: The Danish Non-vitamin K Antagonist Oral Anticoagulation Study. A Cluster Randomized Study Comparing Safety and Efficacy of Edoxaban, Apixaban, Rivaroxaban and Dabigatran for Oral Anticoagulation in Patients With Venous Thromboembolism.
Brief Title: The Danish Non-vitamin K Antagonist Oral Anticoagulation Study in Patients With Venous Thromboembolism (DANNOAC-VTE)
Acronym: DANNOAC-VTE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Gislason, MD,PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DHF2
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Non-vitamin K antagonist oral anticoagulation; Non-vitamin K Antagonist Oral Anticoagulants; Direct-acting Oral Anticoagulants; Novel oral anticoagulant drugs
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Dabigatran; Rivaroxaban; edoxaban; apixaban

STUDY DESIGN:
Intervention Model Description: Cluster randomized cross-over study
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessor will only have a code of each drug and a code for each cluster. Therefore he will not know what drug the clusters have been using. The randomization key will be safely stored at servers at "Statens Serums Institute" (An institute under the Danish Ministry of Health). After the primary and secondary outcome have been evaluated data will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dabigatran (Active Comparator): After randomization, the cluster will use dabigatran to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time.
  Interventions: Drug: Dabigatran Etexilate Oral Capsule; Drug: Rivaroxaban Oral Tablet; Drug: Edoxaban Oral Tablet; Drug: Apixaban Oral Tablet
- Rivaroxaban (Active Comparator): After randomization, the cluster will use rivaroxaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time.
  Interventions: Drug: Dabigatran Etexilate Oral Capsule; Drug: Rivaroxaban Oral Tablet; Drug: Edoxaban Oral Tablet; Drug: Apixaban Oral Tablet
- Edoxaban (Active Comparator): After randomization, the cluster will use edoxaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time.
  Interventions: Drug: Dabigatran Etexilate Oral Capsule; Drug: Rivaroxaban Oral Tablet; Drug: Edoxaban Oral Tablet; Drug: Apixaban Oral Tablet
- Apixaban (Active Comparator): After randomization, the cluster will use apixaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time.
  Interventions: Drug: Dabigatran Etexilate Oral Capsule; Drug: Rivaroxaban Oral Tablet; Drug: Edoxaban Oral Tablet; Drug: Apixaban Oral Tablet

INTERVENTIONS:
Drug: Dabigatran Etexilate Oral Capsule — After cluster randomization, the cluster will use dabigatran to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time. It is the clusters and not the patient that are randomized.
Drug: Rivaroxaban Oral Tablet — After cluster randomization, the cluster will use rivaroxaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time. It is the clusters and not the patient that are randomized.
Drug: Edoxaban Oral Tablet — After cluster randomization, the cluster will use edoxaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time. It is the clusters and not the patient that are randomized.
Drug: Apixaban Oral Tablet — After cluster randomization, the cluster will use apixaban to all their patients with venous thromboembolism when possible for six months. Hereafter the cluster will use the other three NOACs for six months one at the time. It is the clusters and not the patient that are randomized.

SUMMARY:
No randomized head-to-head comparison between the individual Non-vitamin K Antagonist Oral Anticoagulants (NOAC) exists. The DANNOAC-VTE study is a nationwide cluster randomized cross-over study comparing efficacy and safety of the four NOACs, edoxaban, apixaban, rivaroxaban and dabigatran for oral anticoagulation in venous thromboembolism across Danish hospitals.

DETAILED DESCRIPTION:
No randomized head-to-head comparison between the individual Non-vitamin K Antagonist Oral Anticoagulants (NOAC) exists, but such data are warranted to evaluate if the four NOACs are equal in treatment of venous thromboembolism (VTE) without an additional cost of increased bleeding risk. Furthermore, classic randomized trials are highly selective, as elderly and/or fragile patients and patients with comorbidity are underrepresented. Therefore, there is a need of randomized trials that include a broader population of patients.

The DANNOAC-VTE study is a nationwide cluster randomized cross-over study comparing efficacy and safety of the four NOACs, edoxaban, apixaban, rivaroxaban and dabigatran for oral anticoagulation in VTE across Danish hospitals. The aim of the present study is to: 1) examine if the four NOACs are equally effective in treatment of VTE without increasing the risk of major bleeding requiring hospitalization; 2) conduct a randomized study that includes elderly and fragile patients and patients with comorbidity that would otherwise not be included in a traditional randomized clinical trial.

For a variety of reasons, Danish hospitals and clinicians often prefer one particular NOAC. This can make work simpler for the busy clinician, although there may also be economic advantages on a local or a regional larger scale. For a period of two years, this study will replace this individually or hospital preferred selection with a random selection. The hospitals and clinics that participate in this study will be randomly selected to primarily use one specific NOAC for 6 months at a time during a total period of two years. This only applies to patients with VTE that are selected by the physician to be eligible for NOAC treatment. VTE refers to deep vein thrombosis and pulmonary embolism, or a combination of both.

Endpoints

* Primary efficacy outcome: a composite endpoint of new venous thromboembolism or all-cause death.
* Secondary efficacy outcomes: Individually components of the primary endpoints; new venous thromboembolism or all-cause death.
* Primary safety outcome: bleeding requiring hospitalization.
* Other effect measures:

  1. discontinuation of therapy.
  2. adherence to therapy.
  3. other reasons of admission to hospital than included in the primary and secondary endpoint.
* Sensitivity analyses:

  1. primary endpoint stratified by gender.
  2. primary endpoint stratified by age (≤65, 65-75, >75 years of age).
  3. primary endpoint stratified by levels of the CHA2DS2VASc score (0-1, 2-3, >3).
  4. primary endpoint with exclusion of clusters with non-compliance greater than 20% of cluster randomization.
  5. primary endpoint where the actual treatment is used instead of the allocated treatment.
  6. primary safety endpoint stratified by HAS-BLED score.

Information of endpoints and comorbidity is obtained from the Danish National Patient Register based on ICD-10 diagnostic codes and information of vital status and date of death will be obtained from the Central Person Register. Drug discontinuation and adherence will be examined using information from the Danish Registry of Medicinal Product Statistics. The prespecified endpoints will be evaluated after 6 months as intention-to-treat analysis. In addition, the prespecified endpoints will be evaluated after 12 months and 5 years.

A cluster is defined as a hospital or a cardiology clinic. The Clusters will be enrolled in the study from 1. of April 2023 to 1. October 2023.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of VTE in outpatient clinic or as discharge diagnosis after hospitalization.
* A claimed prescription of a NOAC from a Danish pharmacy within 14 days of discharge or outpatient clinic visit.

Exclusion Criteria:

* A prescription of a NOAC within 90 days prior to hospitalization or outpatient clinic visit for VTE.
* Patients with NOAC preference apart from preference consistent with current cluster randomized NOAC.
* Other contraindications mentioned in the "Summary of Product Characteristics" for the respective NOAC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome: a composite endpoint of new venous thromboembolism or all-cause death. | 6 months.
  First occurrence of new venous thromboembolism or all-cause death. Information of endpoints and comorbidity is obtained from the Danish National Patient Register based on ICD-10 diagnostic codes and information of vital status and date of death will be obtained from the Central Person Register. Information of prescribed drug will be obtained using information from the Danish Registry of Medicinal Product Statistics.

SECONDARY OUTCOMES:
Secondary efficacy outcome: New venous thromboembolism. | 6 months.
  Information of endpoints and comorbidity is obtained from the Danish National Patient Register based on ICD-10 diagnostic codes and information of vital status and date of death will be obtained from the Central Person Register. Information of prescribed drug will be obtained using information from the Danish Registry of Medicinal Product Statistics.
Secondary efficacy outcome: All-cause death. | 6 months.
  Information of endpoints and comorbidity is obtained from the Danish National Patient Register based on ICD-10 diagnostic codes and information of vital status and date of death will be obtained from the Central Person Register. Information of prescribed drug will be obtained using information from the Danish Registry of Medicinal Product Statistics.
Primary safety outcome: bleeding requiring hospitalization. | 6 months.
  First occurrence of bleeding requiring hospitalization. Information of endpoints and comorbidity is obtained from the Danish National Patient Register based on ICD-10 diagnostic codes and information of vital status and date of death will be obtained from the Central Person Register. Information of prescribed drug will be obtained using information from the Danish Registry of Medicinal Product Statistics.

OTHER OUTCOMES:
Discontinuation of therapy. | 6 months.
  Drug discontinuation will be examined using information from the Danish Registry of Medicinal Product Statistics.
Adherence to therapy. | 6 months.
  Drug adherence will be examined using information from the Danish Registry of Medicinal Product Statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar H Gislason, MD, PhD, Study Chair — Herlev Gentofte Hospital
Locations (26):
- Denmark (26):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg and Frederiksberg Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen NV
  - Amager Hospital, Copenhagen S
  - Rigshospitalet, Copenhagen Ø
  - Esbjerg Hospital, Esbjerg
  - Nordsjællands Hospital - Frederiksund, Frederikssund
  - Herlev Gentofte Hospital, Gentofte Municipality
  - Glostrup Hospital - Department of Emergency Medicine, Glostrup Municipality
  - Glostrup Hospital - Department of Medicine / Cardiology, Glostrup Municipality
  - Glostrup Hospital - Department of Neurology, Glostrup Municipality
  - Herlev-Gentofte Hospital - Department of Medicine, Herlev
  - Nordsjællands Hospital - Hillerød, Hillerød
  - Hjørring Hospital, Hjørring
  - Holbæk Hospital, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Næstved Hospital, Næstved
  - Odense University Hospital - Department of Cardiology, Odense
  - Odense University Hospital - Department of Emergency Medicine, Odense
  - Odense University Hospital - Department of Geriatrics, Odense
  - Zealand University Hospital - Department of Neurology, Roskilde
  - Zealand University Hospital Roskilde - Department of Cardiology, Roskilde
  - Bornhoms Hospital, Rønne
  - Slagelse Hospital, Slagelse
  - Odense University Hospital Svendborg, Svendborg
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: DANNOAC study webpage — http://dannoac.dk